CLINICAL TRIAL: NCT03750916
Title: Anlotinib Combined With Docetaxel as Second-line Treatment of Patients With Wild-type Advanced Non-squamous NSCLC
Brief Title: Anlotinib Combined With Docetaxel for Advanced Non-squamous Non-Small Cell Lung Cancer
Acronym: ACDFNSNSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L035
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC Anlotinib Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Anlotinib and Docetaxel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride plus Docetaxel (Experimental): Anlotinib(12mg QD PO d1-14, 21 days per cycle) plus Docetaxel (75mg/m2 IV d1) Drug: Anlotinib Hydrochloride plus Docetaxel
  Interventions: Drug: Anlotinib Hydrochloride plus Docetaxel

INTERVENTIONS:
Drug: Anlotinib Hydrochloride plus Docetaxel — Anlotinib Hydrochloride (12mg QD PO d1-14, 21 days per cycle) and Docetaxel (75mg/m2 IV d1)

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore,envisage using anlotinib plus docetaxel treat the advanced Non-squamous non-small cell lung cancer to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This is a multicentre single arm clinical trial conducted in China,the purpose of this study is To Evaluate the Effectiveness and Safety of Anlotinib (12mg QD PO d1-14, 21 days per cycle)Combined with Docetaxel (75mg/m2 IV d1) for advanced Non-squamous non-small cell lung cancer.According to the result of TAX317,the PFS of second line standard chemotherapy was 3 month. Expected the PFS was 5.7. Using PASS11, That calculated the sample size of this study was 41 , according to 10% censoring,the expected sample size is 46.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to patient entry;
* EGFR、ALK mutation-negative；Patients who has failed from the first-line Platinum-based Doublet or single chemotherapy with the advanced non-small cell lung cancer and has not used docetaxel;
* ≥ 18 and ≤ 75 years of age；ECOG PS：0-1;Expected Survival Time: Over 3 months;
* Diagnosed with Non-squamous advanced NSCLC (phase IIIB/IV) through pathology, with measurable nidus(using RECIST 1.1)or recurrent non-squamous non-small cell lung cancer
* Patients who has failed from the first-line Platinum-based Doublet chemotherapy with the advanced non-small cell lung cancer (For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment） Noted: failed from prior treatment means(1) progress disease confirmed by CT; cannot tolerable from standard treatment, such as hematologic toxicities ≥ level 4; non-hematologic toxicities ≥ level 3;damages of heart/liver/kidney ≥ level 2 in CTC AE 4.0;
* Must have at least one measurable lesion as per RECIST 1.1 defined as a lesion that is 10mm in longest diameter imaged by CT scan or MRI；prior topical treatment, such as radiotherapy cryosurgery to the lesions is not allowed in less than 3 months;
* Toxicity caused by prior anti-cancer treatments was restored to ≤ level 1 in CTC AE (4.0),Which accepts the interval of nitrosourea or mitomycin ≥ 6 weeks;Accept other cytotoxic drugs, anti-tumor angiogenesis therapy such as bevacizumab (Avastin), Endo, etc., surgery ≥ 4 weeks;End of radiotherapy (except for local palliative radiotherapy) ≥ 2 weeks;
* The main organs function are normally, the following criteria are met(1)Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L;(2)Biochemical examinations must meet the following criteria: TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.25×ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula);
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped.

Exclusion Criteria:

* Squamous carcinoma(including Adenosquamous carcinoma); Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
* have used Anlotinib、docetaxel before;
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* Medical history and combined history：

  1. Significant brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
  2. The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
  3. Other active malignancies that require simultaneous treatment;
  4. Patients with a history of malignant tumors except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone a curative treatment and have no disease recurrence within 5 years from the start of treatment;
  5. Patients with previous anti-tumor treatment-related adverse reactions (excluding hair loss) who have not recovered to NCI-CTCAE ≤1;
  6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  7. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  8. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  9. Severe acute or chronic infections requiring systemic treatment;
  10. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  11. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
  12. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
  13. Long-term unhealed wounds or fractures;
  14. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  15. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  16. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  17. Events of venous/venous thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
  18. Planned for systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (4 weeks prior to enrollment in other anti-cancer drug clinical trials or within 4 weeks prior to grouping or during the study period Or use mitomycin C) within 6 weeks prior to receiving the test drug. Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before grouping or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks before grouping;
  19. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal medical treatment);
  20. Have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* A known history of HIV testing positive or acquired immunodeficiency syndrome (AIDS);untreated active hepatitis (hepatitis b: HBsAg positive and HBV DNA more than 1 x 103 copy /ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection;
* Serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-11-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Quality of Life score (QoL) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life.